CLINICAL TRIAL: NCT02444234
Title: Steady-State Pharmacokinetics of Tedizolid in Plasma and Sputum of Patients With Cystic Fibrosis
Brief Title: Pharmacokinetics of Tedizolid Phosphate in Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Paul Beringer, Associate Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HS-15-00182
Record Dates: First submitted 2015-05-06; First posted 2015-05-14 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tedizolid PO (Experimental): Tedizolid phophate 200mg tablet
  Interventions: Drug: Tedizolid PO
- Tedizolid IV (Experimental): Tedizolid phophate 200mg IV
  Interventions: Drug: Tedizolid IV

INTERVENTIONS:
Drug: Tedizolid PO — Participants will be randomized to receive tedizolid oral 200mg once daily for 3 days and crossed over to IV after a 1 week washout.
  Arms: Tedizolid PO
Drug: Tedizolid IV — Participants will be randomized to receive tedizolid IV 200mg once daily for 3 days and crossed over to PO after a 1 week washout.
  Arms: Tedizolid IV

SUMMARY:
The proposed study is designed to characterize the pharmacokinetics of intravenous and oral tedizolid in patients with Cystic Fibrosis.

DETAILED DESCRIPTION:
Recent epidemiological studies have demonstrated that the presence of methicillin-resistant Staphylococcus aureus (MRSA) in the airways of patients with CF is associated with more rapid lung function decline and a higher mortality. Tedizolid is a new antibiotic with potent activity against MRSA. Tedizolid is currently FDA approved for treatment of skin soft tissue infections with MRSA. The proposed study is designed to characterize the pharmacokinetics of intravenous and oral tedizolid in patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF based on positive sweat chloride or known CF mutation
* Age > 17 years
* Able to spontaneously expectorate sputum

Exclusion Criteria:

* Any clinically significant laboratory abnormalities
* Presence of an ongoing acute pulmonary exacerbation
* Pregnancy
* Serious past allergy to linezolid or tedizolid
* No alcohol, nicotine, or caffeine-containing products during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a cross-over study where patients with CF received tedizolid 200mg IV or PO once daily for 3 doses followed by a minimum 2 day washout and receipt of the remaining dosage form.
Groups:
- Tedizolid PO/IV: Tedizolid phophate 200mg tablet with crossover to IV
  Tedizolid PO/IV: Participants will be randomized to receive tedizolid oral 200mg once daily for 3 days and crossed over to IV after a minimum 2-day washout.
- Tedizolid IV/PO: Tedizolid phophate 200mg IV with crossover to PO
  Tedizolid IV/PO: Participants will be randomized to receive tedizolid IV 200mg once daily for 3 days and crossed over to PO after a minimum 2-day washout.
Period: First Intervention (3 Days)
Arm/Group | Tedizolid PO/IV | Tedizolid IV/PO
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (2 Day Minimum)
Arm/Group | Tedizolid PO/IV | Tedizolid IV/PO
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention (3 Days)
Arm/Group | Tedizolid PO/IV | Tedizolid IV/PO
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized to receive either tedizolid oral 200 mg tablet or IV 200 mg once daily for 3 days and crossed over to either IV or PO after a minimum of 2 day washout period
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.27 (4.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Creatinine Clearance [Mean (Standard Deviation); unit: mL/min] | 147.6 (32.43)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 21.72 (3.60)

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax)
Description: Cmax was calculated using data collected at 0, 0.5, 1, 2, 3, 4, 8, 24, 48 hours post-dose
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: mg/liter
Groups:
- Tedizolid PO: Tedizolid phophate 200mg tablet with crossover to IV
  Tedizolid PO/IV: Participants will be randomized to receive tedizolid oral 200mg once daily for 3 days and crossed over to IV after a 1 week washout.
- Tedizolid IV: Tedizolid phophate 200mg IV with crossover to PO
  Tedizolid IV/PO: Participants will be randomized to receive tedizolid IV 200mg once daily for 3 days and crossed over to PO after a 1 week washout.
Arm/Group | Tedizolid PO | Tedizolid IV
Number analyzed (Participants) | 11 | 11
mg/liter | 2.22 (0.745) | 2.92 (.624)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Area under the curve was calculated using samples collected at baseline (0 h) , 0.5, 1, 2, 3, 4, 8, 24, and 48 hours post-dose and using the equation AUC=Dose*F/CL
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: mg*h/mL
Arm/Group | Tedizolid PO | Tedizolid IV
Number analyzed (Participants) | 11 | 11
mg*h/mL | 22.1 (5.72) | 20.7 (3.92)

3. Primary Outcome: Time to Peak Plasma Concentration (Tmax)
Description: Tmax was calculated using data collected at 0, 0.5, 1, 2, 3, 4, 8, 24, 48 hours post-dose
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tedizolid PO | Tedizolid IV
Number analyzed (Participants) | 11 | 11
hours | 2.5 (1.33) | 1.36 (0.369)

4. Primary Outcome: Peak Sputum Concentration
Description: Peak sputum concentration was calculated using data collected at 0, 0.5, 1, 2, 3, 4, 8, 24, 48 hours post-dose.
Time Frame: 2 days
Population: One patient could not produce sputum
Measure: Mean (Standard Deviation); unit: mg/liter
Arm/Group | Tedizolid PO | Tedizolid IV
Number analyzed (Participants) | 10 | 10
mg/liter | 1.08 (0.6) | 1.196 (0)

5. Primary Outcome: Area Under the Sputum Concentration Versus Time Curve (AUC)
Description: AUC was calculated using data collected at 0, 0.5, 1, 2, 3, 4, 8, 24, 48 hours post-dose
Time Frame: 2 days
Population: One patient could not produce sputum
Measure: Mean (Standard Deviation); unit: mg*h/mL
Arm/Group | Tedizolid PO | Tedizolid IV
Number analyzed (Participants) | 10 | 10
mg*h/mL | 15.04 (8.92) | 13.53 (7.203)

6. Primary Outcome: Time to Peak Sputum Concentration (Tmax)
Description: Tmax was calculated using data collected at 0, 0.5, 1, 2, 3, 4, 8, 24, 48 hours post-dose. Tmax was derived from pooled sputum data due to sparse samples and therefore do not have standard deviations.
Time Frame: 2 days
Population: One patient could not produce sputum
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Tedizolid PO: Tedizolid phophate 200mg tablet
  Tedizolid PO/IV: Participants will be randomized to receive tedizolid oral 200mg once daily for 3 days and crossed over to IV after a 1 week washout.
- Tedizolid IV: Tedizolid phophate 200mg IV
  Tedizolid IV/PO: Participants will be randomized to receive tedizolid IV 200mg once daily for 3 days and crossed over to PO after a 1 week washout.
Arm/Group | Tedizolid PO | Tedizolid IV
Number analyzed (Participants) | 10 | 10
hours | 4 (0) | 3 (0)

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Tedizolid PO | Tedizolid IV
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tedizolid PO (N=11) | Tedizolid IV (N=11)
Diarrhea (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Observed a large interindividual variability in the absorption rate constant. Due to difficulty of producing sputum, sputum samples were sparse. Did not include a control population to directly compare the pharmacokinetics in CF patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT02444234/Prot_SAP_000.pdf